CLINICAL TRIAL: NCT06863506
Title: Prospective, Multi-cohort, Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of Befotertinib in EGFR-positive Non-classical Mutant Non-small Cell Lung Cancer Patients
Brief Title: Phase II Clinical Study of Befotertinib in EGFR Non-classical Mutant NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown); Hunan Cancer Hospital - the Affiliated Cancer Hospital of Xiangya school of Medicine, Central South University (Unknown); Taizhou Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0190
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G719X, L861Q, or S768I) (Experimental): Patients with EGFR uncommon mutations (G719X, L861Q, or S768I)
  Interventions: Drug: befotertinib
- exon 20 insertion (Experimental): Patients with EGFR exon 20 insertion mutations
  Interventions: Drug: befotertinib

INTERVENTIONS:
Drug: befotertinib — Befotertinib will be administered orally at an initial dose of 75 mg once daily for 21 days, with escalation to 100 mg if tolerated. Treatment continues until disease progression, unacceptable toxicity, or withdrawal.

SUMMARY:
This is a prospective, multi-cohort, single-arm Phase II clinical trial evaluating the efficacy and safety of befotertinib, a third-generation EGFR tyrosine kinase inhibitor (TKI), in patients with advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR non-classical mutations.

The study comprises two independent cohorts:

Cohort 1: Patients with EGFR uncommon mutations (G719X, L861Q, or S768I). Cohort 2: Patients with EGFR exon 20 insertion mutation

Primary endpoint: Objective response rate (ORR) assessed by RECIST 1.1. Secondary endpoints: Disease control rate (DCR), duration of response (DoR), progression-free survival (PFS), overall survival (OS), and safety profile (CTCAE v4.03).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, ECOG performance status 0-2
* Histologically confirmed locally advanced/metastatic NSCLC
* Documented EGFR mutations: Cohort 1 (G719X/L861Q/S768I) or Cohort 2 (exon 20 insertion)
* No prior EGFR-TKI therapy
* Progression or intolerance to ≥1 line of platinum-based chemotherapy -≥1 measurable lesion per RECIST 1.1

Exclusion Criteria:

* Previous EGFR-TKI treatment
* Active CNS metastases (asymptomatic patients with stable lesions allowed)
* Severe cardiovascular disease (e.g., QTc ≥450 ms, myocardial infarction within 6 months)
* Active HBV/HCV/HIV infection
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by RECIST 1.1. | From enrollment until treatment discontinuation (up to 24 months)

SECONDARY OUTCOMES:
progression-free survival (PFS) | From first dose to disease progression or death (assessed up to 36 months)
Disease control rate (DCR) | From enrollment until treatment discontinuation (up to 24 months)
duration of response (DoR) | From the first documented response to disease progression or death, whichever occurs first, assessed up to 36 months.
overall survival（OS） | From enrollment until death from any cause, assessed up to 60 months. Survivors will be censored at the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Li Wen, Prof., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xia Yang, Prof., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang, China